CLINICAL TRIAL: NCT05142332
Title: PROmotion of COvid-19 VA(X)Ccination in the Emergency Department - PROCOVAXED
Acronym: PROCOVAXED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: met interim analysis criteria for early termination
Sponsor: University of California, San Francisco (Other)
Collaborators: Duke University (Other); Thomas Jefferson University (Other); University of Washington (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21-34004; R01AI166967-01 (NIH)
Record Dates: First submitted 2021-11-30; First posted 2021-12-02 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Covid-19 Vaccine; Vaccine Hesitancy
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: Parent Cluster Randomized Trial: Intervention arm is delivery of Covid vaccine messaging Non-intervention arm is usual care. (2 arms)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: PROCOVAXED (Experimental): Covid vaccine educational intervention consisting of vaccine messaging platforms (flyers, videos, scripted face-to-face messaging)
  Interventions: Other: Covid-19 vaccine education materials
- Non-interventional Arm: PROCOVAXED (No Intervention): Usual care

INTERVENTIONS:
Other: Covid-19 vaccine education materials — videos and flyers containing Covid-19 vaccine educational information
  Arms: Intervention Arm: PROCOVAXED

SUMMARY:
The goal of this research is to increase COVID-19 vaccine acceptance and uptake in vulnerable populations whose primary (and often only) health care access occurs in emergency departments (ED Usual Source of Care Patients). Toward this goal, the investigators will conduct one on one interviews and focus groups with ED Usual Source of Care Patients and community partners and produce trusted messaging informational platforms (PROmotion of COvid-19 VA(X)ccination in the Emergency Department - PROCOVAXED) that will address barriers to COVID-19 vaccination, especially vaccine hesitancy. The investigators will then conduct a cluster-randomized, controlled trial of PROCOVAXED platforms in six EDs to determine whether their implementation is associated with greater COVID-19 vaccine acceptance and uptake in ED Usual Source of Care Patients.

DETAILED DESCRIPTION:
The investigator's preliminary work research at 15 ED sites across the US indicates that ED Usual Source of Care patients have particular health care access barriers, needs, and perceptions about vaccines (vaccine hesitancy) that require specific review beyond traditional (non-ED user) community engagement techniques. To gain insight about messaging that effectively addresses these barriers, needs, and perceptions, the investigators will conduct one on one interviews and focus group meetings with ED Usual Source of Care Patients and community partners.

At five safety net EDs (Zuckerberg San Francisco General, Thomas Jefferson University Hospital [Philadelphia], Methodist Hospital [Philadelphia], Harborview Medical Center [Seattle], and Duke University Medical Center [Durham, NC], the investigators will conduct a cluster-randomized, controlled trial of implementation of PROCOVAXED platforms, with COVID-19 and influenza vaccine acceptance rates on post-intervention ED surveys as the primary outcomes. Hypothesis: Implementation of PROCOVAXED platforms in EDs will be associated with increased acceptance of COVID-19 vaccines in ED patients.

One month after subjects' index ED visit enrollment in our PROCOVAXED implementation trial, the investigators will conduct electronic health record review and phone follow-up surveys to determine ED patient uptake (receipt) of COVID-19 vaccines. Hypothesis: Implementation of PROCOVAXED platforms in EDs will be associated with greater COVID-19 vaccine uptake in ED patients.

The investigators will conduct a cluster-randomized, controlled trial (RCT) of implementation of our PROCOVAXED platforms in 5 high-volume, safety net hospital EDs, testing two hypotheses that implementation of PROCOVAXED platforms will be associated with increased acceptance and uptake of COVID-19 vaccines in ED Usual Source of Care Patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years of age) patients who are receiving care at participating Emergency Departments and have not yet received a COVID-19 vaccine (PROCOVAXED)

Exclusion Criteria:

* major trauma patients
* patients transferred from another hospital, chronic care facility, nursing home or hospice,
* patients unable to participate in an interview because of intoxication, altered mental status or critical illness
* incarcerated patients
* patients on psychiatric holds
* patients who have received a COVID-19 vaccine
* under suspicion for acute COVID-19 illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rodriguez, MD, Principal Investigator — University of California, San Francisco
Locations (7):
- United States (7):
  - San Francisco General Hospital Emergency Department, San Francisco, California
  - University of California, San Francisco - Parnassus, San Francisco, California
  - Duke University Hospital, Durham, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Jefferson Methodist Hospital, Philadelphia, Pennsylvania
  - University of Washington-Harborview Emergency Department, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez RM, Nichol G, Eucker SA, Chang AM, O'Laughlin KN, Pauley A, Rising KL, Eswaran V, Morse D, Li C, Patel A, Duber HC, Arreguin M, Shughart L, Glidden D; PROCOVAXED Study Network. Effect of COVID-19 Vaccine Messaging Platforms in Emergency Departments on Vaccine Acceptance and Uptake: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2023 Feb 1;183(2):115-123. doi: 10.1001/jamainternmed.2022.5909. PMID 36574256
- [Derived] Gentsch AT, Butler J, O'Laughlin K, Eucker SA, Chang A, Duber H, Geyer RE, Guth A, Kanzaria HK, Pauley A, Rising KL, Chavez CL, Tupetz A, Rodriguez RM. Perspectives of COVID-19 vaccine-hesitant emergency department patients to inform messaging platforms to promote vaccine uptake. Acad Emerg Med. 2023 Jan;30(1):32-39. doi: 10.1111/acem.14620. Epub 2022 Nov 22. PMID 36310395
- [Derived] Rodriguez RM, O'Laughlin K, Eucker SA, Chang AM, Rising KL, Nichol G, Pauley A, Kanzaria H, Gentsch AT, Li C, Duber H, Butler J, Eswaran V, Glidden D. PROmotion of COvid-19 VA(X)ccination in the Emergency Department-PROCOVAXED: study protocol for a cluster randomized controlled trial. Trials. 2022 Apr 21;23(1):332. doi: 10.1186/s13063-022-06285-x. PMID 35449064

RESULTS

PARTICIPANT FLOW:
Groups:
- Zuckerberg San Francisco Hospital; University of California San Francisco Hospital -Parnassus; Thomas Jefferson University Hospital; University of Washington-Harborview Emergency Department: First Condition: Control
- Duke University Hospital; Jefferson Torresdale Hospital; Jefferson Methodist Hospital: First condition: Intervention
Period: Overall Study
Arm/Group | Zuckerberg San Francisco Hospital | University of California San Francisco Hospital -Parnassus | Duke University Hospital | Thomas Jefferson University Hospital | Jefferson Torresdale Hospital | Jefferson Methodist Hospital | University of Washington-Harborview Emergency Department
Started (Participant came in on the day site was randomized to this condition and participant was consented) | 166 | 27 | 110 | 97 | 12 | 12 | 117
Received PROCOVAXED Intervention | 82 | 8 | 49 | 27 | 2 | 3 | 50
C C Control | 79 | 18 | 52 | 61 | 9 | 4 | 52
Completed | 161 | 26 | 101 | 88 | 11 | 7 | 102
Not Completed | 5 | 1 | 9 | 9 | 1 | 5 | 15
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0 | 0 | 2 | 6
Not completed — Left ED | 3 | 0 | 4 | 6 | 1 | 2 | 6
Not completed — Physician Decision | 0 | 0 | 2 | 1 | 0 | 0 | 3
Not completed — Became ineligible (e.g. developed altered mental status) | 2 | 0 | 1 | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm: PROCOVAXED | Non-interventional Arm: PROCOVAXED | Total
Number analyzed (Participants) | 221 | 275 | 496
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [31 to 53] | 39 [29 to 54] | 39 [30 to 54]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 86 | 119 | 205
  Male | 134 | 155 | 289
  Other | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants could answer more than one race or ethnicity
  Participants
    African American | 71 | 122 | 193
    American Indian or Alaskan Native | 14 | 4 | 18
    Asian | 5 | 7 | 12
    Latinx | 50 | 47 | 97
    Native Hawaiian or Pacific Islander | 4 | 6 | 10
    White, non-Latinx | 85 | 98 | 183
    Other | 23 | 25 | 48
Region of Enrollment [Number; unit: participants]
  United States | 221 | 275 | 496
Has a primary care clinic or physician [Count of Participants; unit: Participants]
  Yes | 119 | 158 | 277
  No | 101 | 117 | 218
  Unsure | 1 | 0 | 1
Primary language [Count of Participants; unit: Participants]
  English | 196 | 239 | 435
  Spanish | 22 | 25 | 47
  Other | 3 | 11 | 14
Housing status [Count of Participants; unit: Participants]
  Housed | 172 | 236 | 408
  Marginal | 10 | 9 | 19
  Unhoused | 38 | 30 | 68
  No answer given | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Covid-19 Vaccine Acceptance in the Emergency Department: PROCOVAXED
Description: Participant acceptance of the COVID-19 vaccine assessed by the question "Would you accept the COVID-19 vaccine in the emergency department today if your doctor or provider asked you to get it?" The response choices for this question are "Yes", "No", and "No, but I might consider getting it at some other time".
  This question will be asked once at the end of the Emergency Department visit.
Time Frame: Within 6 hours of intervention
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm: PROCOVAXED | Non-interventional Arm: PROCOVAXED
Number analyzed (Participants) | 221 | 275
Participants | 57 | 33
Statistical Analysis 1: Comparison: Intervention Arm: PROCOVAXED vs Non-interventional Arm: PROCOVAXED; Test type: Superiority; p < 0.001, Regression, Logistic; Adjusted absolute difference = 11.9, 95% CI 2-sided [4.5 to 19.3]

2. Primary Outcome: Covid-19 Vaccine Uptake: PROCOVAXED
Description: Participation uptake of the COVID-19 vaccine 30 days after enrollment assessed by confirmation of receipt of vaccine in one of 3 ways:
  1. Receipt in emergency department during index (enrollment) visit
  2. Electronic health record review 30 days after index visit
  3. Follow up phone call to participant at 28 to 30 days - We are asking patients if they received a COVID-19 vaccine since their index emergency department visit.
Time Frame: Within 30 days of intervention
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm: PROCOVAXED | Non-interventional Arm: PROCOVAXED
Number analyzed (Participants) | 221 | 275
Participants | 44 | 24
Statistical Analysis 1: Comparison: Intervention Arm: PROCOVAXED vs Non-interventional Arm: PROCOVAXED; Test type: Superiority; p < 0.001, Regression, Logistic; Adjusted absolute difference = 7.9, 95% CI 2-sided [1.7 to 14.1]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Intervention Arm: PROCOVAXED | Non-interventional Arm: PROCOVAXED
All-Cause Mortality (participants affected / at risk) | 0/221 | 0/275
Serious Adverse Events (participants affected / at risk) | 0/221 | 0/275
Other Adverse Events (participants affected / at risk) | 0/221 | 0/275

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT05142332/Prot_SAP_001.pdf